CLINICAL TRIAL: NCT00791115
Title: Salvage Prostatectomy After Radiotherapy: Whole-Mount Histopathological Validation for Tumor-Targeted Salvage HDR Brachytherapy
Brief Title: Salvage Prostatectomy After Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0350-CE; NIH CA12156
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; prostatectomy; radiotherapy; prostatectomy after radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- prostatectomy after radiotherapy (Experimental)
  Interventions: Procedure: whole-mount sectioning of the prostate

INTERVENTIONS:
Procedure: whole-mount sectioning of the prostate — A standard open retropubic radical prostatectomy will be performed. Whole fresh prostate is be embedded in gel and oriented in the anatomic position in a plastic cylinder using wood skewers. Standard pathology reports are generated from this tissue

SUMMARY:
The purpose of this study is to compare the location of the cancer found in the prostate gland after it is removed to the location that was predicted on the MRI scan during biopsy. In this way, we can better determine if the Magnetic Resonance Imaging (MRI) was accurate, and if the MRI could be safely used to guide other types of treatments such as brachytherapy. We also plan to carefully measure how frequently surgery is able to completely remove the cancer, as well as the side effects and effectiveness of surgery after radiotherapy. The study will be coordinated and closely integrated with a separate concurrent study of MRI-guided prostate biopsy, which will be performed prior to accrual to this trial (UHN 05-0641-C).

DETAILED DESCRIPTION:
Two hundred and nineteen thousand new cases of prostate cancer have been projected in the Unites States for 2007, with external beam radiotherapy (EBRT) constituting the mainstay of local therapy for an increasing proportion of newly diagnosed patients. Despite improvements in the delivery and reduction in associated toxicity of external beam radiotherapy, local persistence or recurrence of disease remains prevalent in 25-51% of patients. Local disease after EBRT is a risk factor for subsequent metastatic progression and prostate cancer-specific mortality, and is a cause of morbidity including hematuria, obstructive uropathy, and chronic pain. Given its prevalence, and the lack of satisfactory local salvage treatments, fear of prostate cancer recurrence has been shown to impose a substantial burden of suffering in patients.

Stereotactic needle placement under MRI-guidance enables two critical steps in tumor-targeted brachytherapy: 1) directly guiding brachytherapy catheters to sites of tumor recurrence, and 2) permitting treatment planning and delivery to be based on 3D MRI images. MRI-based HDR brachytherapy will precisely identify the location of brachytherapy catheters relative to the target volumes and adjacent normal structures at risk of radiation injury, obviating the need for invasive saturation (24-100) mapping biopsies.

This study will build the evidence supporting the concept of tumor-targeted salvage HDR brachytherapy, by providing further histopathological validation of the method.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment of UHN 05-0641-C
* Histological evidence of cancer on MRI-guided prostate biopsy
* PSA doubling time > 6 months
* ECOG 0 or 1
* All patients must give written informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed

Exclusion Criteria:

* Contraindications to salvage prostatectomy
* Previous rectal surgery for IBD or cancer such that an ileo-anal anastomosis is present.
* Radiological evidence of regional or distant metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-06; Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
To Validate virtual dosimetry plans for tumor-targeted salvage (High-Dose-Rate) HDR brachytherapy against co-registered whole-mount prostatectomy specimens. | Patients will have follow-up assessments at 1,3 and 6 months and 1,2,3 and 5 years after surgery.

SECONDARY OUTCOMES:
Preliminary evaluation of surgical margin status, toxicity and QOL, and biochemical control after salvage RP. | Patients will have follow-up assessments at 1,3 and 6 months and 1,2,3 and 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ménard, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada